CLINICAL TRIAL: NCT04898153
Title: First-in-Human (FIH) Study of the Xeltis Hemodialysis Access Graft (aXess)
Brief Title: First-in-Human (FIH) Study of the Xeltis Hemodialysis Access Graft
Acronym: aXess-FIH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-08
Record Dates: First submitted 2021-04-13; First posted 2021-05-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: End Stage Renal Disease; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aXess (Experimental): Patients will be implanted with the Xeltis hemodialysis access graft (aXess)
  Interventions: Device: aXess

INTERVENTIONS:
Device: aXess — Patients will be implanted with one Xeltis hemodialysis access device (aXess) in the arm

SUMMARY:
A feasibility study is to assess the preliminary safety and performance of the Xeltis hemodialysis access (aXess) graft.

DETAILED DESCRIPTION:
A prospective, single arm, non-randomized FIH feasibility study to evaluate the preliminary safety and performance of the Xeltis hemodialysis access graft in subjects older than 18 years with end-stage renal disease, who plan to undergo hemodialysis for at least the first 6 months after study access creation, and are deemed not suitable for fistula creation by the operating surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years with end-stage renal disease (ESRD) who are not, or who are no longer, candidates for creation of an autogenous AV fistula, and therefore require placement of an AV graft in the upper extremity to start or maintain hemodialysis therapy
* Suitable anatomy for the implantation of an aXess graft
* The patient has been informed about the nature of the study, agrees to its provisions, and has provided written informed consent
* The patient has been informed and agrees to pre- and post- procedure follow up
* Life expectancy of at least 12 months

Exclusion Criteria:

* History or evidence of severe cardiac disease (NHYA Functional Class IV and/or EF <30%), myocardial infarction within six months of study entry, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* Stroke within six months before study entry
* Active clinically significant autoimmune / inflammatory disease, immunodeficiency (including AIDS / HIV), use of immunosuppressive therapy or medication that likely interferes with restorative therapies
* Abnormal blood values (e.g. leurkopenia with white blood cell (WBC) count < 4,000/mm3 and/or anemia with hemoglobin <8g/dL and/or thrombocytopenia < 100,000/mm3) that could influence patient recovery and/or graft hemostasis
* Any active local or systemic infection (WBC > 15,000/mm3)
* Uncontrolled or poorly controlled diabetes (hemoglovin A1c > 8% despite standard care) or hospitalization for poor glucose control within the previous 6 months
* Reduced liver function, defined as: >2x the upper limit of normal for serum bilirubin, aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase; International Normalized Ratio (INR) > 1.5 or prothrombin time (PT) > 18 seconds
* Known heparin-induced thrombocytopenia
* Active bleeding disorder and/or any coagulopathy or thrombo embolic disease
* History or evidence of severe peripheral vascular disease in the upper limbs
* Known or suspected central vein obstruction on the side of planned graft implantation
* Previous dialysis access graft in the operative limb unless the aXess graft can be placed more proximally than the previous failed graft
* More than 1 failed dialysis access graft in the operative limb
* Anticipated renal transplant within 6 months
* Subjects receiving a forearm graft which crosses the elbow
* Allergies to study device (Nitinol) or agents/medication, such as contrast agents, aspirin, or clopidogrel, that cant be controlled medically
* Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives
* Subject is participating in another study
* Previous enrollment in this study
* Any other condition which, in the judgement of the investigator would preclude adequate evaluation for the safety and efficacy of the study conduit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from device related serious adverse events | 6 months
  The number of patients who have a device related serious adverse event
Functional patency of graft | 6 months
  The number of patients with a functionally patent graft

SECONDARY OUTCOMES:
Freedom from device related serious adverse events | 12, 18, 24, and 60 months
  The number of patients who have a device related serious adverse event
Functional patency of graft | 12, 18, 24, and 60 months
  The number of patients with a functionally patent graft
Patency (primary, primary assisted, and secondary) of graft | 6, 12, 18, 24, and 60 months
  The number of patients with a patient graft
Time to potential central venous catheter removal | Assessed retrospectively at 30 days
  Time that patients with a central venous catheter could have had the catheter removed after the Xeltis hemodialysis access graft was placed
Time to loss of patency (primary, primary assisted, and secondary) | 6, 12, 18, 24, and 60 months
  Number of days from implant to graft occlusion in patients who no longer have a patent graft
Rate of access related interventions required to achieve/maintain patency | 6, 12, and 24 months
  Number of interventions that were performed on grafts to achieve/maintain patency
Rate of access site infections | 6, 12, and 24 months
  Number of access graft sites that become infected
Proportion of hemodialysis (HD) sessions completed via central venous catheter | 12 months
  Number of hemodialysis sessions performed with a central venous catheter vs. the number of sessions performed with the Xeltis hemodialysis access graft
Number of days with central venous catheter in place (catheter contact time) | 12 months
  Number of days the patients have a central venous catheter in place irrespective of access abandonment
Pseudoaneurysm formation | 6, 12, and 24 months
  Number of grafts that have a pseudoaneurysm form

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vermassen, MD, Principal Investigator — UZ Ghent
Locations (6):
- Belgium (3):
  - A.Z. Sint Jan, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Ghent, Ghent
- Universita degli studi dell'Insubria, Varese, Italy
- P. Stradins Clinical University Hospital, Riga, Latvia
- Vilnius University Hospital Santaros Klinikos Corpus A., Vilnius, Lithuania

REFERENCES:
- [Derived] Tozzi M, De Letter J, Krievins D, Jushinskis J, D'Haeninck A, Rucinskas K, Miglinas M, Baltrunas T, Nauwelaers S, Schoen FJ, Virmani R, De Vriese AS, Moll F, Vermassen F. Endogenous tissue restoration in a hemodialysis conduit: Performance and safety after 1-year of follow-up. J Vasc Access. 2025 Nov 21:11297298251395823. doi: 10.1177/11297298251395823. Online ahead of print. PMID 41272425